CLINICAL TRIAL: NCT06338722
Title: Evaluation of the Making it Work Program for Systemic Sclerosis
Brief Title: Making it Work Program for Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-397
Record Dates: First submitted 2024-02-09; First posted 2024-04-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Scleroderma, Systemic
Keywords: work
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Intervention receives the Making it work program Wait list Control receives usual care but will be offered the program after the intervention groups finish
Masking Description: People will know what group they are in when they are invited to attend the intervention sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Complete questionnaires Attend one 2 hour weekly virtual meeting for 5 weeks and an individual meeting with an occupational therapist and with a vocational counselor
  Interventions: Other: Making it Work Systemic Sclerosis
- control group (No Intervention): Complete questionnaires

INTERVENTIONS:
Other: Making it Work Systemic Sclerosis — One 2 hour virtual meeting per week for 5 weeks, plus an individual meeting with an occupational therapist and a vocational counselor
  Arms: Intervention group

SUMMARY:
The purpose of this clinical trial is to see if an online intervention program for people with Systemic Sclerosis (scleroderma) helps keep people in the workforce and increase self-confidence in dealing with challenges at work. The program is called Making it Work Systemic Sclerosis.

Researchers will compare a group who gets the program to a group who will get the program at a later point in time (wait list control group) to see if self-confidence in dealing with work challenge gets better.

People in the Making it Work group will complete questionnaires and attend one 2 hour meetings each week for 5 weeks and meet with an occupational therapist and vocational counselor. People in the wait list control group will complete the questionnaires and participate in the program at a later point in time.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed (full-time, part-time)
* Over 18 and less than or equal to 67 years of age
* Reside and work in the United States
* Self-report diagnosis with systemic sclerosis (scleroderma; systemic sclerosis)
* Report concerns about risk for job loss
* Possess sufficient spoken English to participate in a group
* Have device with audio and visual videoconferencing capabilities
* Be willing to participate in a 2.0 hour virtual meeting once a week for 5 weeks
* Be willing to complete assigned pre-meeting worksheets
* Be willing to meet virtually with both an occupational therapist and vocational counselor after the 5th weekly sessin.

Exclusion Criteria:

* Not working (full-time, part-time, self-employed, contract work)
* Pregnant
* Less than 18 and over 67 years of age
* Do not work in the United States
* Do not report are not concerned about job loss
* Do not have a device with audio and visual videoconferencing capabilities
* Do note communicate sufficiently in English
* Are not able to participate in the program for 5 weeks
* Are not wiling to complete pre-meeting worksheets
* Not willing to meet with both an occupational therapist and vocational counselor.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Job Related Self-efficacy Scale | baseline, 5 weeks, 12 weeks, 24 weeks
  Measures self-efficacy for managing problems/challenges at work
Job Self-Efficacy Scale | baseline, 5 weeks, 12 weeks, 24 weeks
  Measures confidence in concepts targeted by the Making it Work Program such as disease management at work, stress management, ability to communicate effectively, obtaining job accommodations

SECONDARY OUTCOMES:
Work Productivity and Activity Impairment Questionnaire Specific Health Problem Subscale | baseline, 5 weeks, 12 weeks, 24 weeks
  Measures absenteeism [secondary outcome; hours and days missed from work due to SSc] and presenteeism [secondary outcome; at-work productivity].
The Work Instability Scale | baseline, 5 weeks, 12 weeks, 24 weeks
  Measures risk for future work loss

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Poole, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States